CLINICAL TRIAL: NCT04414241
Title: Hydroxychloroquine to Prevent SARS-CoV-2 Infection Among Healthcare Workers: Randomized Controlled, Open-label, Phase 3 Clinical Trial
Brief Title: Hydroxychloroquine to Prevent SARS-CoV-2 Infection/COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202087; 20923 (Other: OGITT-INS)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2020-06

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2 infection; Hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine prophylaxis plus standard measures of personal protection.
  Interventions: Drug: Hydroxychloroquine
- Control (No Intervention): Standard measures of personal protection.

INTERVENTIONS:
Drug: Hydroxychloroquine — A loading dose of 600mg of hydroxychloroquine orally on the first day, followed by 400mg of hydroxychloroquine orally every-other-day and use of standard measures of personal protection provided from the hospital for 8 weeks.
  Arms: Hydroxychloroquine

SUMMARY:
The purpose of this study is to determine whether hydroxychloroquine is an effective prophylactic regimen to prevent SARS-CoV-2 infection among healthcare workers. Participants will be randomized into two parallel groups. The first arm will evaluate the use of hydroxychloroquine every-other-day plus standard measures of protection for the prevention of SARS-CoV-2. The second arm will evaluate the use of standard measures of protection for the prevention of SARS-CoV-2. The target enrollment is 320 participants. Each study participant will be monitored for SARS-CoV-2 seroconversion in weekly visits or for the development of COVID-19 symptoms for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare workers in service during the COVID-19 outbreak including medical, nurse, technical, and auxiliary staff.
2. Negative rapid serologic and molecular testing for SARS-CoV-2.
3. Written informed consent.

Exclusion Criteria:

1. Presents COVID-19 symptoms including cough, fever, myalgias, headaches, loss of smell, and taste.
2. Prior (last 30 days), current or planned use (during study period) of hydroxychloroquine, chloroquine sulfate, or azithromycin.
3. Known cardiac disease or a history of prolonged QT syndrome.
4. Known allergy or intolerance to hydroxychloroquine and/or chloroquine sulfate.
5. Use of concomitant medications that are contraindicated with the use of hydroxychloroquine.
6. Other reported medical conditions, such as glucose-6-phosphate dehydrogenase deficiency, hepatic or renal insufficiency, or visual acuity or field disturbances, that make study participation not in the individual's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Efficacy: Proportion of participants with positive molecular or serologic testing for SARS-CoV-2 | Eight weeks
Safety: Proportion of participants with grade 3 or more adverse events | Eight weeks

SECONDARY OUTCOMES:
Tolerability: Proportion of participants that discontinue prophylactic treatment due to grade 1 or 2 adverse events | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Llanos, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia; Eduardo Gotuzzo, MD, Study Chair — Universidad Peruana Cayetano Heredia; Max Grogl, PhD, Study Chair — U.S. Naval Medical Research Unit Six; Patricia García, MD, MPH, PhD, Study Chair — Universidad Peruana Cayetano Heredia; Manuel Espinoza, MD, Study Chair — Instituto de Nacional de Salud
Locations (3):
- Peru (3):
  - Centro Médico Naval "Cirujano Mayor Santiago Távara", Callao
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Cayetano Heredia, Lima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Llanos-Cuentas A, Schwalb A, Quintana JL, Delfin B, Alvarez F, Ugarte-Gil C, Guerra Gronerth RI, Lucchetti A, Grogl M, Gotuzzo E. Hydroxychloroquine to prevent SARS-CoV-2 infection among healthcare workers: early termination of a phase 3, randomised, open-label, controlled clinical trial. BMC Res Notes. 2023 Feb 28;16(1):22. doi: 10.1186/s13104-023-06281-7. PMID 36849996